CLINICAL TRIAL: NCT04507373
Title: 7T Magnetic Resonance Spectroscopy and Skeletal Muscle Biopsy Findings in Statin
Brief Title: 7T Magnetic Resonance Spectroscopy and Skeletal Muscle Biopsy Findings in Statin Associated Adverse Muscle Events
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: No grant obtained. Enrolled participants were not assigned to the intervention and was study terminated
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, Zahid Ahmad, Associate Professor, University of Texas Southwestern Medical Center
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Basic Science
Other Study IDs: STU 072016-015
Record Dates: First submitted 2019-01-31; First posted 2020-08-11 (Actual); Results first posted 2023-02-14 (Actual); Last update posted 2023-02-14 (Actual); Status verified 2023-01

CONDITIONS: Muscle Cramp; Ache; Weakness, Muscle; Statin Adverse Reaction
MeSH Terms: conditions — Muscle Cramp; Pain; Muscle Weakness | interventions — Simvastatin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: Double Blind
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Placebo (Placebo Comparator): Following the baseline period, subject will be randomized to receive either simvastatin or an identical placebo at a dose of 40 mg/day for a period of 10 weeks.
  Interventions: Drug: Simvastatin 40mg
- Simvastatin 40mg (Active Comparator): Following the baseline period, subject will be randomized to receive either simvastatin or an identical placebo at a dose of 40 mg/day for a period of 10 weeks.
  Interventions: Drug: Simvastatin 40mg

INTERVENTIONS:
Drug: Simvastatin 40mg — 40mg oral daily for 10 weeks

SUMMARY:
Over 40 million Americans take statins to reduce their risk of atherosclerotic cardiovascular disease (ASCVD). Unfortunately, 10 to 20% stop taking them due to statin-associated muscle symptoms (e.g. pain, aches, weakness, cramps, or stiffness) (1, 2). The pathophysiology of these statin-associated muscle symptoms (SAMS) has remained elusive. Consequently, no objective diagnostic method exists, causing confusion for patient and providers since muscle symptoms can often be multifactorial.

DETAILED DESCRIPTION:
The overall objectives of this project are to identify the underlying cause of SAMS and establish an in-vivo imaging technique to detect SAMS. The central hypothesis of this pro-posal is that statins directly inhibit mitochondrial function in SAMS patients. Our rationale is based on our own preliminary data indicating that simvastatin - the most common statin to cause SAMS - can directly inhibit oxidative phosphorylation (OXPHOS) in mice. Since such changes can be detected in vivo in humans utilizing 31P magnetic resonance spectroscopy (MRS) techniques, the investigators will use a state-of-the art 7 Tesla (7T) MRS instrument to study the so-leus muscles of SAMS patients. Additionally, the investigators will validate the MRS findings by doing func-tional studies in muscle biopsy specimens.

The investigators propose double-blind randomized, placebo-controlled pilot study in 15 SAMS pa-tients and 15 controls. Study participants will be treated with simvastatin 40 mg daily or place-bo for 10 weeks. The investigators will perform 7T MRS of soleus muscles at randomization and either at first complaint of muscle symptoms or at the end of 10 weeks if no muscle symptoms occur, whichever occurs first. Quadriceps muscle biopsies will also be done immediately following the second MRS scan.

ELIGIBILITY:
Inclusion

• Adults, age > 18 ys or < 80 yrs. Patients reporting complaints of statin-associated muscle symptoms, aches, weakness, cramps, or stiffness in the legs.

Exclusion Criteria

* Patient who drink large quantities of grapefruit juice (> 1 quart daily).
* Patients on the following drugs for which the FDA has issued restrictions for using simvastatin 40 mg daily do to an increased risk of severe muscle injury such as itraconazole, posaconazole, ketoconazole, erythromycin, clarithromycin, telithromycin, HIV-1 protease inhibitors, nefazodone, gemfibrozil, cyclosporine, danazol, amiodarone, amlodipine, ranolazine, and verapamil.
* Patients with muscle-related pain that is not related to statin-use (e.g. muscle aches from strain or trauma) or remains unexplained.
* Any patients with underlying non-statin related muscle disorders.
* Presence of any clinically significant uncontrolled endocrine disease known to influence serum lipids or lipoproteins.
* Conditions of severe acute vascular stress (acute coronary syndrome, ischemic stroke, or major vascular surgery) within prior 3 months.
* Any patients with a history of severe or life-threatening reactions to statins including rhabdomyolysis (defined as evidence of organ damage with CK >10,000 IU/L), CK elevation > 10 times the upper limit of normal, cognitive decline, transaminitis, or allergic reactions.
* History of fibromyalgia or rheumatologic disease with symptoms that may be confounded with statin-related muscle complaints.
* Patients unable to maintain their current activity level or planning to increase their activity level (e.g. new exercise regimen). Such changes may have acute effects on muscle metabolism.
* Pregnant or breast-feeding women. Statins are teratogenic, and the effects of high magnetic fields on a fetus are unknown.
* Women of reproductive age not on effective contraception. Adequate contraceptive measures include intrauterine device (IUD); bilateral tubal ligation; condom or diaphragm plus either contraceptive sponge, foam or jelly.
* Any person with implanted metal, because of MRS safety.
* Use of any active investigational drugs within 1 month or 5 half-lives, whichever is longer.
* History of antibodies to HMGCoA.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2018-08-17 (Actual); Primary Completion 2021-12-20 (Actual); Study Completion 2021-12-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Zahid Ahmad, M.D., Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- UT Southwestern Medical Center, Dallas, Texas, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The 3 participants who were consented/ enrolled were not assigned/ randomized to the interventions because no grant was obtained for the study to continue further and the study was terminated.
Period: Overall Study
Arm/Group | Placebo | Simvastatin 40mg
Started | 0 | 0
Completed | 0 | 0
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: The 3 participants who were consented/ enrolled were not assigned/ randomized to the interventions because no grant was obtained for the study to continue further and the study was terminated.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Simvastatin 40mg | Total
Number analyzed (Participants) | 0 | 0 | 0
Age, Categorical
Age, Continuous
Sex: Female, Male
Race (NIH/OMB)

OUTCOME MEASURES:

1. Primary Outcome: The Mitochondrial Changes In Muscles During Statin Use
Description: Study participants being treated with Simvastatin 40mg daily, or placebo for 10 weeks. Investigators will isolate mitochondrial from muscle biopsy sample and compare mitochondrial oxygen consumption rates, ultrastructural changes, and gene expression
Time Frame: 10 weeks
Population: The participants who were consented/ enrolled were not assigned/ randomized to the interventions because no grant was obtained for the study to continue further and the study was terminated.
Arm/Group | Placebo | Simvastatin 40mg
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Data was never collected
Description: Data was never collected
Arm/Group | Placebo | Simvastatin 40mg
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2018-04-25): https://cdn.clinicaltrials.gov/large-docs/73/NCT04507373/Prot_000.pdf
  • Statistical Analysis Plan (2016-07-07): https://cdn.clinicaltrials.gov/large-docs/73/NCT04507373/SAP_001.pdf